CLINICAL TRIAL: NCT04416607
Title: Ovarian Response to Controlled Ovarian Stimulation Measured Through the Follicular Output Rate (FORT)
Brief Title: Corifollitropin Alpha and Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87020518800005327
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- corifollitropin alpha (Experimental): Ovarian stimulation protocol is performed with a single dose of 100 μg (<60 kg) or 150 μg (≥60 kg) of corifollitropin alpha (Elonva, Schering-Plough, Brazil), plus gonadotropin-releasing hormone antagonist co-treatment (Ganirelix 25 mcg/day, Orgalutran, Schering-Plough, Brazil) in a flexible protocol (at least 1 follicle >14 mm or 3 or more follicles >12 mm).
  Interventions: Drug: Corifollitropin Alfa
- menotropin (Active Comparator): 150-300 IU/day HMG (menotropin, Menopur, Ferring, Brazil) is administered, starting on cycle day 3, according to age, AMH level and AFC, plus gonadotropin-releasing hormone antagonist co-treatment (Ganirelix 25 mcg/day, Orgalutran, Schering-Plough, Brazil) in a flexible protocol (at least 1 follicle >14 mm or 3 or more follicles >12 mm).
  Interventions: Drug: Menotropins

INTERVENTIONS:
Drug: Corifollitropin Alfa — Primary outcome measure is ovarian response measured by FORT. Drugs are administrated for controlled ovarian stimulation prior in vitro fertilization.
  Other Names: Elonva® (Schering-Plough)
  Arms: corifollitropin alpha
Drug: Menotropins — Primary outcome measure is ovarian response measured by FORT. Drugs are administrated for controlled ovarian stimulation prior in vitro fertilization.
  Other Names: Menopur® (Ferring)
  Arms: menotropin

SUMMARY:
Objective: To study whether an administration of corifollitropin alpha modifies the follicular cohort, measured by Follicular Output Rate (FORT), compared to human menopausal gonadotropin (HMG), in infertile patients undergoing in vitro fertilisation (IVF).

M/M: 306 infertile patients undergoing in vitro fertilisation (IVF). Ovarian stimulation protocol will be performed with a single dose of 100 μg (<60kg) or 150 μg (≥60kg) corifollitropin alpha in group 1 (n=147), and 150-300 IU/day human menopausal gonadotropin (HMG) according to age, antimullerian hormone (AMH) level and antral follicle count (AFC) in group 2 (n=150).

Moreover, FORT will be calculated as the ratio of pre-ovulatory follicle (16-22 mm in diameter) count on day of HCG×100/small antral follicle (3-8 mm) count at baseline.

DETAILED DESCRIPTION:
Patients will be allocated for convenience into two groups: those who would receive corifollitropin alpha (Group 1) or HMG (Group 2).

Ovarian stimulation protocol will be performed with a single dose of 100 μg (<60 kg) or 150 μg (≥60 kg) of corifollitropin alpha (Elonva, Schering-Plough, Brazil) in group 1, which could be followed by daily administration of HMG beginning on day 8 if necessary; in group 2 150-300 IU/day HMG (menotropin, Menopur, Ferring, Brazil) will be administered, starting on cycle day 3, according to age, AMH level and AFC, plus gonadotropin-releasing hormone antagonist co-treatment (Ganirelix 25 mcg/day, Orgalutran, Schering-Plough, Brazil) in a flexible protocol (at least 1 follicle >14 mm or 3 or more follicles >12 mm). Doses will be adjusted as needed by the patient according to the ultrasound, which is performed with a 6 MHz multifrequency transvaginal probe (Toshiba, Japan). The criterion for HCG administration (5.000 IU Choriomon, Biopharma, Brazil) will be at least three follicles greater than 17 mm, and then, 36 hours later, transvaginal oocyte retrieval was performed. After 3 or 5 days, one or two good-quality embryos will be transferred. It will be performed intracytoplasmic sperm injection (ICSI) instead of conventional IVF when major male factor is presented.

Primary outcome measure is FORT. Secondary outcome measures include number of oocytes retrieved, MII, duration of stimulation, number of embryos, embryo quality and clinical pregnancy rate. Adverse events, such as ovarian hyperstimulation syndrome (OHSS) or drug-related complications are also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles;
* Body mass index (BMI) of <33.0 kg/m².

Exclusion Criteria:

* Previous ovarian surgery;
* Current diagnosis of polycystic ovarian syndrome (PCOS) or other endocrinopathies;
* History of autoimmune or metabolic disorders.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
FORT | 15 days
  FORT is calculated as the ratio of pre-ovulatory follicle (16-22 mm in diameter) count on day of HCG × 100/small antral follicle (3 -8 mm in diameter) count at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joao Sabino Lahorgue da Cunha Filho, Ph.D., Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Centro de Reproduçao Humana Insemine, Porto Alegre, RGS
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, RGS

IPD SHARING:
Plan to Share IPD: No